CLINICAL TRIAL: NCT03733015
Title: Can Daily Sessions of rTMS to the Left DLPFC Boost Diffuse Noxious Inhibitory Control and Pain Thresholds in Healthy Subjects
Brief Title: Daily Sessions of rTMS to the Left DLPFC Modulate the Pain Thresholds and CPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 54271916.8.0000.0068
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Pain Relief
Keywords: repetitive transcranial magnetic stimulation; dorsolateral prefrontal cortex; pain thresholds
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS group (Active Comparator): Transcranial magnetic stimulation (TMS) is used to stimulate small regions of the brain. During a TMS procedure, a magnetic field generator, or "coil", is placed near the head of the person receiving the treatment. TBS refers to a rTMS protocol where pulses are applied in bursts of three, delivered at a frequency of 50 Hz and an inter-burst interval of 200 ms (5 Hz).
  Interventions: Device: repetitive transcranial magnetic stimulation
- High frequenct rTMS group (Active Comparator): High frequency refers to a rTMS protocol where pulses are applied in at 10Hz frequency
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Repetitive transcranial Magnetic Stimulation (rTMS) can be used to temporary modify the brain activity.

SUMMARY:
The main purpose of the study is to assess whether repeated sessions of repetitive trancranial magnetic stimulation (rTMS) applied on left dorsolateral prefrontal cortex main boost the pain thresholds.

DETAILED DESCRIPTION:
Pain is the largest health-related burden on society and, despite many decades of pain research, there are still few effective treatments. Since pain experience is a construct of the central nervous system (CNS), chronic pain has been recently thought to be a CNS disorder.

Repetitive transcranial magnetic stimulation (rTMS) is a safe, non-invasive technique for cerebral cortex stimulation and the clinical applications of which have expanded considerably in recent years. Recent studies have been shown that 'classical' rTMS to different cortical areas temporary reduce chronic and acute pain, suggesting that rTMS may ´have some clinical application in future management of chronic pain. However, new rTMS paradigms involving theta burst stimulation (TBS) have recently been described with the major clinical advantage to be much shorter than 'classical' rTMS. The investigators hypothesize that cTBS would yield analgesic effects similar to or, possibly, even stronger than those produced by 'classical' rTMS. The investigators will carry out a sham-controlled, randomized, double-blind, crossover study in healthy volunteers, to compare the analgesic effects of two rTMS protocols over dorsolateral prefrontal cortex: classical high-frequency rTMS (10 Hz), and TBS. As rTMS-induced analgesia may be dependent on changes in pain modulatory systems, the investigators will analyze the effects of the stimulation on conditioned pain modulation (CPM). More specifically, the investigators will compare the effects of multiple sessions of rTMS on the inhibition of a test experimental stimulus induced by heterotopic noxious stimuli, to assess possible changes in diffuse noxious inhibitory controls.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Major medical conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Pressure pain thresholds (PPT) | The study comprises two interventions of four experimental sessions on consecutive days (Day-1 to Day-4). Changes from Day-1 at Day-4 will be investigated.
  Pressure will be applied at a rate of 30 kPa/s perpendicularly to the surface of the skin using a handheld algometer (1-cm2 probe; Somedic, Hörby, Sweden). Three readings at the pressure pain threshold (PPT) will be made at 1-minute intervals, at four sites; i) right elbow, ii) left elbow, iii) right leg and iv) left leg. The data will be reported in kPa.
Cold pain thresholds, heat pain thresholds and supra-thresholds painful stimuli | The study comprises two interventions of four experimental sessions on consecutive days (Day-1 to Day-4). Changes from Day-1 at Day-4 will be investigated.
  The temperature of the thermode is slowly decreased or increased to the maximum tolerable levels. The participant will click a button as soon as the tolerable level has been reached, which will bring the temperature back to baseline 32 degrees Celsius. Thresholds are determined by raising or dropping the temperature slowly from baseline skin temperature until the participant reports feeling of pain. The experimenter will then determine the temperature that is consistently rated as moderately painful by applying a temperature above the threshold level and asking the participant to rate the pain from 0 (no pain) to 10 (most intense pain imaginable).
Condition pain modulation (supra-thresholds painful stimuli ): visual analogue scale (VAS: 0-100mm) | The study comprises two interventions of four experimental sessions on consecutive days (Day-1 to Day-4). Changes from Day-1 at Day-4 will be investigated.
  First, the volunteers will immerse the left hand in a bucket with water and ice at 4° C for around 45-60 seconds to reach a VAS pain of 60-70/100mm. Immediately after, supra-thresholds painful stimuli over the right leg will be repeated in a randomized order. The supra-thresholds painful stimuli will be reported in a VAS scale (from 0 to 10).
Condition pain modulation (pressure pain thresholds): visual analogue scale (VAS: 0-100mm) | The study comprises two interventions of four experimental sessions on consecutive days (Day-1 to Day-4). Changes from Day-1 at Day-4 will be investigated.
  First, the volunteers will immerse the left hand in a bucket with water and ice at 4° C for around 45-60 seconds to reach a VAS pain of 60-70/100mm. Immediately after, pressure pain thresholds over the right leg will be repeated. The pressure pain thresholds will be reported in kPa.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Enrico De Martino, Aalborg, North Denmark
  - Enrico De Martino, Aalborg

IPD SHARING:
Plan to Share IPD: No